CLINICAL TRIAL: NCT02383667
Title: Clinical Comparison of Electrocardiograms Collected Using an Ambulatory Holter
Acronym: Orbital
Status: Completed | Type: Observational
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Sponsor
Organization: University of Toledo (Other)
Other Study IDs: Orbital
Record Dates: First submitted 2015-03-03; First posted 2015-03-09 (Estimated); Results first posted 2019-10-07 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-09

CONDITIONS: Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Electrocardiograms: Any patient within the hospital either for procedure or for admission will be screened. Patients will be simultaneously be hooked up to two ambulatory Holter monitors for the period of time to be not less than one hour.
  One holter will use standard electrodes in a standard electrode distribution. The second holter will use dry electrodes in a derived; data will be collected for 1-6 hours. After the data is collected the Holters will be removed and the data will be downloaded into the reading software to be scanned.
  Interventions: Device: Electrocardiogram holter

INTERVENTIONS:
Device: Electrocardiogram holter

SUMMARY:
The objective of the study is to compare electrocardiograms using ambulatory holter monitor with dry electrodes in a harness versus using an ambulatory holter with standard sticky electrodes (Red Dot) on monitored patients within the hospital. Patients will be simultaneously be hooked up to two ambulatory Holter monitors for the period of time to be not less than one hour. One holter will use standard electrodes in a standard electrode distribution. The second holter will use dry electrodes in a derived.

ELIGIBILITY:
Inclusion Criteria:

* Any patient within the hospital either for procedure or for admission

Exclusion Criteria:

* Patients who cannot wear a Holter monitor
* Patients undergoing an MRI or have other contraindications for wearing an ambulatory Holter monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients within the hospital either for a procedure or for admission
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Cummings, MD, Principal Investigator — The University of Toledo
Locations (1):
- University of Toledo, Health Science Campus, Toledo, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment was done in the hospital setting with patients that were admitted. start of enrollment was 3/26/2013-3/9/15.
Groups:
- Patients With Electrocardiograms: Any patient within the hospital either for procedure or for admission will be screened. Patients will be simultaneously be hooked up to two ambulatory Holter monitors for the period of time to be not less than one hour.
  One holter will use standard electrodes in a standard electrode distribution. The second holter will use dry electrodes in a derived; data will be collected for 1-6 hours. After the data is collected the Holters will be removed and the data will be downloaded into the reading software to be scanned.
  Electrocardiogram holter
Period: Overall Study
Arm/Group | Patients With Electrocardiograms
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Electrocardiograms
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 16
Age, Continuous [Mean (Full Range); unit: years] | 74.6 [40 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Arrythmia
Description: quality of data obtained between harness and holter.
  Subjective evaluation:
  -Quality of the data will be rated on a 0 - 10 scale with 0 being unreadable and 10 being excellent
Time Frame: 15 minutes
Population: there were 13 females and 7 males, mean age of 74.65
Measure: Mean (Standard Deviation); unit: Quality rating
Arm/Group | Patients With Electrocardiograms
Number analyzed (Participants) | 20
Quality rating
  harness | 4.6 (2.30332)
  holter | 7.95 (1.877715)

ADVERSE EVENTS:
Arm/Group | Patients With Electrocardiograms
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes